CLINICAL TRIAL: NCT02879513
Title: A Randomized Phase III Trial of Comparing Combination Administration of Paclitaxel and Cisplatin Versus CEF as Adjuvant Chemotherapy in Breast Cancer Patients With Pathological Partial Response and Complete Response to Neoadjuvant Chemotherapy
Brief Title: Trial of Adjuvant Chemotherapy in Breast Cancer Patients With Pathological Partial Response and Complete Response to Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Lu, Director of Department of Breast Surgery, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RenJiH-BC-003
Record Dates: First submitted 2016-07-17; First posted 2016-08-25 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2019-03

CONDITIONS: Invasive Ductal Breast Cancer; Tubular Breast Cancer; Mucinous Breast Cancer; Inflammatory Breast Cancer
MeSH Terms: conditions — Carcinoma, Ductal, Breast; Inflammatory Breast Neoplasms | interventions — Paclitaxel; Cisplatin; Epirubicin; Cyclophosphamide; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Switch to CEF (Active Comparator): Epirubicin 75 mg/m² IV push on day 1 every 3 weeks for 4 cycles. Cyclophosphamide 500 mg/m² IV push on day 1 every 3 weeks. 5-fluoruracil 500 mg/m² IV push on day 1 every 3 weeks.
  Interventions: Drug: Epirubicin; Drug: Cyclophosphamide; Drug: 5-fluoruracil
- Continue the neoadjuvant regimen (Experimental): Paclitaxel: 80 mg/m² i.v. given weekly on day 1 q day 8 for 16 weeks. Cisplatin: 25 mg/m² weekly on day 1 ,8,and 15 q day 28 for 4 cycles.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin
- Pathological complete response group with chemotherapy (Experimental): Paclitaxel: 80 mg/m² i.v. given weekly on day 1 q day 8 for 16 weeks. Cisplatin: 25 mg/m² weekly on day 1 ,8,and 15 q day 28 for 4 cycles.
  Interventions: Drug: Paclitaxel; Drug: Cisplatin
- Pathological complete response group with no chemotherapy (No Intervention)

INTERVENTIONS:
Drug: Paclitaxel
  Other Names: Taxol
  Arms: Continue the neoadjuvant regimen; Pathological complete response group with chemotherapy
Drug: Cisplatin
  Arms: Continue the neoadjuvant regimen; Pathological complete response group with chemotherapy
Drug: Epirubicin
  Arms: Switch to CEF
Drug: Cyclophosphamide
  Arms: Switch to CEF
Drug: 5-fluoruracil
  Other Names: 5-FU
  Arms: Switch to CEF

SUMMARY:
This trial will compare the administration of 2 cycles of paclitaxel and cisplatin (DP) versus 4 cycles of CEF as adjuvant chemotherapy for the patients with locally advanced breast cancer and who were pathological partial response to DP as neoadjuvant chemotherapy. Those who had pathological complete response to DP will be randomized to have 2 cycles of DP or have no further chemotherapy.

DETAILED DESCRIPTION:
All the patients who had neoadjuvant chemotherapy and had pathological complete response (pCR) or partial response to DP will enrolled in this trial. Those who had pCR will randmized to have two cycles of DP as adjuvant chemotherapy or have no further chemotherapy. Those patients who had PR will be randomized to have two cycles of DP or four cycles of CEF. All the patients with hormonal receptor positive or Her2 overexpress tumors are allowed to accept endocrine therapy or anti-Her2 target therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥18years and ≤70 years;
2. Patients with locally advanced breast caner and had weekly paclitaxel and cisplatin as neoadjuvant chemotherapy.
3. Patients with pathological partial response or pathological complete response to neoadjuvant chemotherapy according to the Response Evaluation Criteria in Solid Tumors (RECIST).
4. Endocrine therapy and trastuzumab were allowed to use.
5. ECOG 0-2;
6. Adequate bone marrow function:WBC≥4.0×109/L, Absolute neutrophil count（ANC）≥1.5×109/L, Platelets（PLT）≥100×109/L, Hemoglobin（Hb）≥90g/L;aspartate aminotransferase(AST),Alanine aminotransferase (ALT)≤1.5 upper normal limit (UNL), creatinine≤1.5 UNL, bilirubin≤1.5UNL;
7. No obvious main organs dysfunction.

Exclusion Criteria:

1. Unwilling or unable to use an acceptable method of contraception in 8 weeks (including 8 weeks) after final dose of test drug;
2. Patient is pregnant or breast feeding;
3. Metastatic breast cancer;
4. Any evidence of sense or motor nerve disorders;
5. Patients with medical conditions taht indicate intolerant to neoadjuvant therapy, including uncontrolled cardiovascular disease, severe infection;
6. Any concurrent malignancy other than breast cancer;
7. Know severe hypersensitivity to any drugs in this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2014-01; Primary Completion 2020-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Up to 5 years

SECONDARY OUTCOMES:
overall survival (OS) | Up to 5 years
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 4 months during adjuvant therapy
regional recurrence free survival (RRFS) | 5 years
local recurrence free survival (LRFS) | 5 years
distant-disease- free survival (DDFS) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiaotong University School of Medicine, Renji Hospital, Shanghai, Shanghai Municipality, China